CLINICAL TRIAL: NCT06207617
Title: Evaluation of Soft and Hard Tissue Dimensional Changes Following Immediate Implant Placement in Molar Extraction Sockets With or Without Bone Graft: A Randomized Controlled Clinical Trial
Brief Title: Dimensional Changes Following Immediate Implant Placement in Molar Extraction Sockets With or Without Bone Graft
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Misr International University (Other)
Responsible Party: Principal Investigator, Ahmed Abo El Futtouh, Ahmed Aboulfettouh, Misr International University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IDCE.N9
Record Dates: First submitted 2023-12-17; First posted 2024-01-17 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Immediate Implants

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate implant placement + customized healing abutment (Experimental): After atraumatic extraction, flapless immediate implant of a suitable size will be placed using sequential drills of the Straumann implant system for osteotomy preparation. According to the prosthetically driven planned position, implant will be placed. Primary stability of the implant will be measured by rotational insertion torque, to be more than or equal 30 Ncm. All patients will receive an immediate anatomical customized healing abutment fabricated by adding flowable composite to the temporary cylindrical abutment mimicking the shape of the socket at the marginal gingiva, then it will be screwed to the implant.
  Interventions: Procedure: Immediate implant placement + customized healing abutment
- Immediate implant placement + xenogeneic bone graft material + customized healing abutment (Active Comparator): After atraumatic extraction, immediate implant will be placed as mentioned-above, then particulate xenogeneic bone graft will be packed into the gap between the implant and the buccal plate mesially and distally. bone grafting will be up to the level of the buccal bone crest, followed by screwing the customized healing abutment.
  Interventions: Procedure: Immediate implant placement + xenogeneic bone graft material + customized healing abutment

INTERVENTIONS:
Procedure: Immediate implant placement + customized healing abutment — Immediate implant placement in fresh extraction molar sites + customized healing abutment fabricated by adding flowable composite to the temporary cylindrical abutment mimicking the shape of the socket at the marginal gingiva, then it will be screwed to the implant. no grafting material included in this arm
  Other Names: IIP+customized healing abutment
  Arms: Immediate implant placement + customized healing abutment
Procedure: Immediate implant placement + xenogeneic bone graft material + customized healing abutment — Immediate implant placement in fresh extraction molar sites + xenogenic bone graft + customized healing abutment fabricated by adding flowable composite to the temporary cylindrical abutment mimicking the shape of the socket at the marginal gingiva, then it will be screwed to the implant.
  Arms: Immediate implant placement + xenogeneic bone graft material + customized healing abutment

SUMMARY:
Statement of problem: The majority of studies on immediate implant placement are related to the maxillary esthetic zone. Literature concerning Immediate implant placement in the posterior region is scarce. Furthermore, there is paucity of evidence on alveolar bone dimensional changes following immediate implant placement in fresh extraction sockets of posterior teeth. Adding to that, negligible evidence is known about the soft tissue alterations which take place during modeling and remodeling phases of socket healing process; regarding the molar sites. Nevertheless, Immediate installation into a molar socket raises an extra challenge for the clinicians, because of the different anatomical features of the extraction sockets compared to that of the single-rooted teeth in the anterior zone. In addition to, implant positioning difficulties; due to the amount of the residual inter-radicular bone after extraction. Aim of the study: To assess the bucco-lingual ridge collapse after immediate implant placement in lower 1st molar sites either with customized healing abutment only; or with xenogeneic bone graft and customized healing abutment. Materials and methods: The current study will include 28 non-restorable lower 1st molar teeth indicated for extraction in the posterior area. Patients will randomly be assigned into two equal groups: the test group; Immediate implant placement + customized healing abutment group and the control group; Immediate implant placement +bone graft+ customized healing abutment group. The presented trial will investigate the following outcomes: bucco-lingual ridge collapse as the primary outcome, together with mid-facial recession, total volume gain/loss, buccal soft tissue contour, bucco-lingual bone width, and vertical bone changes as the secondary outcomes after 12 months

DETAILED DESCRIPTION:
After administration of local anesthesia, flapless atraumatic extraction will be performed using peristomes inserted along the root surface, apical pressure and rocking motion will be applied circumferentially to cut the periodontal ligaments. After initial luxation using Harpoon luxators, bayonet forceps will be used to deliver the tooth out of the socket. Often separation of the mesial and distal roots will be employed, to facilitate tooth delivery without impinging the soft and hard tissue architecture. Socket debridement will be done using socket curette and saline irrigation, to make sure the socket is thoroughly clean with no remnants of any periapical pathosis.

Immediate implant placement + customized healing abutment (Test group): After atraumatic extraction, flapless immediate implant of a suitable size will be placed using sequential drills of the Straumann implant system for osteotomy preparation. According to the prosthetically driven planned position, implant will be placed. Primary stability of the implant will be measured by rotational insertion torque, to be more than or equal 30 Ncm. All patients will receive an immediate anatomical customized healing abutment fabricated by adding flowable composite to the temporary cylindrical abutment mimicking the shape of the socket at the marginal gingiva, then it will be screwed to the implant.

Immediate implant placement + xenogeneic bone graft material + customized healing abutment (Control) After atraumatic extraction, immediate implant will be placed as mentioned-above, then particulate xenogeneic bone graft will be packed into the gap between the implant and the buccal plate mesially and distally. bone grafting will be up to the level of the buccal bone crest, followed by screwing the customized healing abutment.

Objectives:

* To compare Bucco-lingual ridge dimension between the two groups at baseline and one-year postoperative.
* To compare the volumetric changes in the labial soft tissue contour between the two groups assessed in mm and mm3.
* To assess and compare the Bucco-palatal bone width, and vertical bone changes in mm using cone beam computed tomography (CBCT) preoperative and at 12 Months.
* To evaluate mid facial gingival recession assessed in mm by the volumetric analysis.
* To assess peri-implant soft tissue parameters by plaque and bleeding indices.
* To assess any surgical or prosthetic complications.
* To assess Implant Failure and Implant Survival Rate

ELIGIBILITY:
Inclusion Criteria:

* Adults from the age of 18 - 50 years of both genders.
* Patients with non-restorable single bounded mandibular 1st molar tooth indicated for extraction.
* Periodontally healthy patients with good oral hygiene.
* Intact interradicular bone with 2-3 mm width, assessed by CBCT.
* Thin buccal plate of bone (1 mm or less) among both of the mesial and distal root, assessed by CBCT.
* Intact gingival tissue with at least 2 mm keratinized tissue.
* Patients accepts to provide written informed consent.

Exclusion Criteria:

* Molar sites indicated for extraction with roots of close proximity to vital structures as inferior alveolar nerve.
* Pregnant females.
* Smokers as smoking is a contraindication for any plastic periodontal surgery (Khuller, 2009).
* Handicapped and mentally retarded patients.
* Patients undergoing chemotherapy and/or radiotherapy.
* Presence of systemic disease that would affect wound healing.
* Presence of active infection with soft tissue communication.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Bucco-lingual ridge dimension | 12 months
  volumetric analysis software will calculate the overall labio-palatal ridge width (mm)

SECONDARY OUTCOMES:
total buccal volume loss (mm3) | 12 months
  volumetric analysis software will calculate the overall labio-palatal ridge width (mm)
Horizontal labio-palatal bone width | 12 months
  A reference line will be constructed along the palatal surface of the implant on the cross-sectional cut of the postoperative CBCT volume. Then, both initial (T0) and postoperative (T1) CBCT volumes will be superimposed on the fusion module. The horizontal labio-palatal width will be measured from the reference line to the outer labial bone at three levels below the labial bone crest: 0mm, 2mm and 5mm at T0 and T1. The difference between T1 and T0 will be calculated and compared to record the mm and % horizontal labio-palatal bone collapse.
Vertical crestal bone level changes | 12 months
  a horizontal line will be placed to mark the crestal labial bone on both the initial and postoperative CBCT volumes separately. Then, both initial and postoperative CBCT volumes will be superimposed on the fusion module. A vertical linear measurement perpendicular to both lines will be done to record the mm vertical crestal bone level changes.
mid-facial recession | 12 months
  using a volumetric analysis software
linear volumetric change of buccal soft tissue contour | 12 months
  at 2, 4, 6mm below the free gingival margin (FGM) at baseline, 6-and 12-months postoperative. using a volumetric analysis software

IPD SHARING:
Plan to Share IPD: No